CLINICAL TRIAL: NCT02587897
Title: Sonographic Tissue Morphology in Early Stage Work-related Median Nerve Pathology
Brief Title: Musculoskeletal Health of the Upper Extremity in Emerging Health Professionals
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency); Loma Linda University (Other); National Center for Dental Hygiene Research and Practice (Other)
Responsible Party: Principal Investigator, Shawn Roll, Associate Professor, University of Southern California
Other Study IDs: HS-15-00004; 1R01OH010665-01A1 (NIH)
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2023-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Ultrasonography; Nerve Conduction Velocity; Ergonomics; Work Related Injury; Cumulative Trauma Disorders
MeSH Terms: conditions — Carpal Tunnel Syndrome; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Dental Hygiene Students: Students enrolled in the 2-year dental hygiene academic coursework programs at the University of Southern California and Loma Linda University who are exposed to high-intensity work-related hand activities as part of their training program.
  Interventions: Other: Academic Coursework; Other: Work-Related Hand Activities
- Occupational Therapy Students: Students enrolled in the 2-year occupational therapy academic coursework program at the University of Southern California.
  Interventions: Other: Academic Coursework

INTERVENTIONS:
Other: Academic Coursework — Didactic training provided by the university through coursework and laboratory training that meets requirements of the accreditation standards provided by the professional society associated with each professional degree granting program.
Other: Work-Related Hand Activities — Exposure to intensive training in the use of dental scaling tools as part of laboratory courses, as well as fieldwork and residency training during the academic degree program.
  Groups: Dental Hygiene Students

SUMMARY:
Carpal tunnel syndrome is the most expensive upper extremity work-related musculoskeletal disorder, impacting 10 million people annually and costing employers up to $113,695 per incident. There is currently no established method to detect this disorder prior to the onset of symptoms and nerve damage. Preliminary research suggests that sonography-a relatively inexpensive, widely available, increasingly portable technology-can provide a non-invasive and pain-free method of early detection that could reduce incidence, improve targeted interventions and ultimately reduce costs. The primary aims of this study are to establish predictive validity of a novel method for early detection using sonographic imaging and to identify task components of intensive functional hand activity associated with morphologic changes.

DETAILED DESCRIPTION:
This longitudinal study will follow dental hygiene students-a high-risk population with minimal retrospective and controlled prospective task exposure-for two years and compare them to a non-exposed cohort of occupational therapy students to investigate the primary aims. This research is directed at the National Occupational Research Agenda's (NORA) Healthcare and Social Assistance sector with a focus on the National Institute of Occupational Safety and Health's (NIOSH) Exposure Assessment and Musculoskeletal Disorders cross-sectors. Intermediate outcomes of this research will establish sonographic imaging as an early detection tool for workplace-screening and inform methods for combining measures of nerve morphology, neurophysiology, and subjective symptoms for predicting the development of work-related carpal tunnel syndrome. This work will also inform the development of targeted preventive interventions for task components of intensive hand activities that are related to changes in tissue morphology. Identifying morphologic changes in early-stages of pathology and the specific task components linked to these changes are the first steps toward early detection and prevention of work-related carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in one of the academic programs (i.e., register and pay for classes)

Exclusion Criteria:

* <18 years of age
* Prior carpal tunnel release surgery
* Prior diagnosis of median nerve pathology or other poly-neuropathy that includes the median nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll a total of 120 dental hygiene students from the University of Southern California (USC) and Loma Linda University (LLU), as well as 60 occupational therapy students from USC.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Symptom & Function Reports on the Boston Carpal Tunnel Questionnaire at 2 years | Baseline and 2 years

SECONDARY OUTCOMES:
Change from Baseline in Cross-Sectional Area of Median Nerve in the Carpal Tunnel Measured with Sonography at 1 year | Baseline and 1 year
Change from Baseline in Cross-Sectional Area of Median Nerve in the Carpal Tunnel Measured with Sonography at 2 years | Baseline and 2 years
Change from Baseline in Vascularity within the Median Nerve Measured with Doppler Sonography at 1 year | Baseline and 1 year
Change from Baseline in Vascularity within the Median Nerve Measured with Doppler Sonography at 2 years | Baseline and 2 years
Change from Baseline in Nerve Conduction Velocity of the Median Nerve at 1 year | Baseline and 1 year
  Nerve conduction velocity testing of the median nerve includes physiological measurement of the ability of the nerve to conduct electrical signals using nerve conduction testing equipment (Sierra Wave) with a surface stimulator at the wrist and surface electrodes on the second and fifth digits.
Change from Baseline in Nerve Conduction Velocity of the Median Nerve at 2 years | Baseline and 2 years
  Nerve conduction velocity testing of the median nerve includes physiological measurement of the ability of the nerve to conduct electrical signals using nerve conduction testing equipment (Sierra Wave) with a surface stimulator at the wrist and surface electrodes on the second and fifth digits.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn C Roll, PhD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Loma Linda Univeristy Dental Hygiene Program, Loma Linda, California
  - USC Musculsokeletal Sonography & Occupational Performance Laboratory, Los Angeles, California
  - USC Dental Hygiene, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
Once manuscripts from the project become available, datasets used to produce manuscripts will be shared with individual peers under the auspices of the PI. Only de-identified data in final databases, will be shared; raw data will not be shared. Data from secondary analyses beyond the specific aims will only be shared under the auspices of the investigators involved. When authorized, data will be made available to requestors under a data-sharing agreement that provides for: (1) using the data for research only, (2) securing the data using appropriate techniques, (3) destroying or returning the data after analyses are completed, and (4) providing the PI with a summary of how the data were used. Requestors agree to protect the intellectual property rights of the PI, or other investigators as indicted, by appropriately acknowledging the source of the data in any document or presentation, which may include oversight or authorship on work that is based substantially on the shared data.

REFERENCES:
- [Background] Yao B, Evans KD, Roll SC. Assessing the Potential for Error in Investigating Intraneural Vascularity: A Need for a Standardized Imaging Protocol. J Diagn Med Sonogr. 2023 Nov;39(6):549-559. doi: 10.1177/87564793231193396. PMID 38074490
- [Background] Fang Y, Kapellusch JM, Baker NA, Roll SC. CHARACTERIZING PHYSICAL STRAIN IN NON-ROUTINIZED CLINICAL WORK THROUGH OBSERVATION: AN EXAMPLE OF ORAL HEALTHCARE PROVIDERS. Proc Int Symp Hum Factors Ergon Healthc. 2024 Sep;13(1):134-139. doi: 10.1177/2327857924131015. PMID 39430719
- [Background] Loomis KJ, Roll SC. External wrist ratio is not a proxy for internal carpal tunnel shape: Implications for evaluating carpal tunnel syndrome risk. Clin Anat. 2024 Nov;37(8):869-877. doi: 10.1002/ca.24132. Epub 2024 Jan 3. PMID 38173294
- [Background] Grutzmacher I, Schicht R, Schlaeger R, Sill V. [Hemodynamics of pulmonary circulation in patients with chronic obstructive lung disease and pulmonary hypertension as dependent on the theophylline concentration of the serum]. Prax Klin Pneumol. 1984 Jan;38(1):19-25. No abstract available. German. PMID 6709589
- [Background] Sloan H. J. Maxwell Chamberlain, 1906-1968. Ann Thorac Surg. 1981 Aug;32(2):109-10. doi: 10.1016/s0003-4975(10)61016-8. No abstract available. PMID 7020616
- [Background] Fotter R, Hollwarth M. [Water syphon test and gastro-oesophageal reflux during childhood (correlation with the clinical findings and oesophageal manometry) ]. Rofo. 1981 Jul;135(1):53-6. doi: 10.1055/s-2008-1056830. German. PMID 6214479
- [Background] A WHO Meeting. Prevention of hepatocellular carcinoma by immunization. A WHO meeting. Bull World Health Organ. 1983;61(5):731-44. PMID 6317213
- [Background] Pozzi F, Sousa CO, Plummer HA, Andrade B, Awokuse D, Kono N, Mack WJ, Roll SC, Michener LA. Development of shoulder pain with job-related repetitive load: mechanisms of tendon pathology and anxiety. J Shoulder Elbow Surg. 2022 Feb;31(2):225-234. doi: 10.1016/j.jse.2021.09.007. Epub 2021 Oct 14. PMID 34656782
- [Background] Yao B, Roll SC. An ultrasound study of the mobility of the median nerve during composite finger movement in the healthy young wrist. Muscle Nerve. 2022 Jan;65(1):82-88. doi: 10.1002/mus.27437. Epub 2021 Oct 27. PMID 34648193
- [Background] Yao B, Takata SC, Mack WJ, Roll SC. Modeling extracurricular activity participation with physical and mental health in college students over time. J Am Coll Health. 2023 May-Jun;71(4):1232-1240. doi: 10.1080/07448481.2021.1926263. Epub 2021 Jul 9. PMID 34242536
- [Background] Roll SC, Hardison ME, Forrest JL, Colclazier NL, Sumi JY, Baker NA. A standardized protocol for the comprehensive assessment of dental hygiene work. Work. 2021;69(3):1041-1052. doi: 10.3233/WOR-213534. PMID 34219697
- [Background] Fang Y, Tung KD, Beleno-Sanchez J, Forrest JL, Roll SC. Characterization of Tasks and Time Efficiency of Dental Hygiene Students During Clinical Training. J Dent Hyg. 2020 Oct;94(5):30-37. PMID 33008947
- [Background] Roll SC, Takata SC, Yao B, Kysh L, Mack WJ. Sonographic reference values for median nerve cross-sectional area: A meta-analysis of data from healthy individuals. J Diagn Med Sonogr. 2023 Sep;39(5):492-506. doi: 10.1177/87564793231176009. Epub 2023 Jun 6. PMID 37654772